CLINICAL TRIAL: NCT07269444
Title: Efficacy of IPACK Block Combined With Intra-articular Steroid Injection in Advanced Knee Osteoarthritis: A Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Collaborators: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Halil Ibrahim Altun, Director, Head of pain medicine, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: knee osteoarthritis
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis (Knee OA); IPACK Block Multimodal Analgesia; Intraarticular Injection; Ultrasound Guided Injection
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Comparison of the Effectiveness of Ultrasonography-Guided Intra-Articular Steroid Injection and IPAC

SUMMARY:
Osteoarthritis is the insufficiency of joint cartilage resulting from the interaction of genetic, metabolic, and biochemical factors, and is accompanied by secondary inflammation. This condition is a pathological process involving the interactive damage and repair of cartilage, bone, and synovium. Osteoarthritis is the most common joint disease worldwide and causes the greatest physical disability. The most prominent symptom is pain. It typically increases with activity and decreases with rest. As the disease progresses, the pain becomes more pronounced with lighter activity, eventually occurring at rest and at night.

The knee joint is a synovial joint formed between the femoral condyles and the tibia. Sensory innervation of the knee joint is provided by branches of the femoral, obturator, and sciatic nerves. Pain from knee osteoarthritis is a common problem that can cause disability and impair quality of life. In many patients with chronic knee pain due to osteoarthritis, pharmacological methods and/or physical therapy may not provide adequate analgesia. Knee arthroplasty is the most frequently used treatment option for advanced knee osteoarthritis. However, it is sometimes not applicable due to patient comorbidities. The most commonly used interventional method for analgesia in knee osteoarthritis today is intra-joint steroid injection. This slows inflammation in the cartilage and can prevent osteophyte formation. However, frequent steroid injections can lead to both short-term pain relief and osteoporosis in the bone.

In recent years, different alternatives for the treatment of osteoarthritis-related knee pain have become prominent. The nerves that provide pain sensation to the knee joint originate from both the anterior and posterior sides. The IPACK block, a simple, practical method performed under ultrasound guidance, is often thought to block the area innervating the posterior knee, but cadaver studies suggest that the anterior geniculate nerves are also blocked. This can be an alternative treatment option for additional analgesia in patients with advanced knee osteoarthritis.The aim of this study is to investigate the effects of IPACK block combined with steroid injection into the knee joint on pain scores in painful patients diagnosed with chronic knee osteoarthritis.

DETAILED DESCRIPTION:
Patients presenting to the Algology Outpatient Clinic of Istanbul Cemil Taşçıoğlu City Hospital between January 2024 and September 2025 with knee pain and diagnosed with stage 3-4 knee osteoarthritis based on clinical, radiological, and laboratory tests were scheduled for the procedure. The procedure was performed on only one knee; the second knee was not treated.

On the morning of the procedure, patients' NRS-11 and WOMAC scores were recorded. After being taken to the operating room, patients were placed in the supine position. Electrocardiography, pulse oximetry, and non-invasive blood pressure monitoring were performed. Intravenous access was established. The painful knee area was prepared and draped in a sterile manner using povidone-iodine-based solution. Ultrasonography (US) was used to image the knee joint and its surrounding area. In patients undergoing knee steroid administration (IASI), a 22-gauge, 90-mm needle was advanced from the suprapatellar area to the joint space under ultrasound guidance. The joint capsule was punctured, and 40 mg of triamcinolone acetonide was injected into the joint.

Patients undergoing IASI+IPACK (infiltration of the space between the popliteal artery and the posterior knee capsule) block were placed in the supine position, in accordance with monitoring and sterilization guidelines. Following the same procedure as described above, the knee was first IASI performed, and a pillow was placed under the knee at 30 degrees of flexion. After imaging the knee joint space with an US-guided medial approach, the probe was advanced approximately 2-3 cm above the patella level, starting from the distal medial epicondyle of the femur. Then, 15 ml of 0.25% bupivacaine + 4 mg dexamethasone mixture was administered between the joint capsule and the popliteal artery and vein, where the femoral condyles end and the femoral body begins, using a 22-gauge 90 mm needle.

After the procedure, patients were observed in our inpatient ward for at least 2 hours to monitor for potential side effects. One week after the injection, all patients were given an exercise booklet to follow their rehabilitation program at home.

Patients were advised to use 500 mg of paracetamol (up to four tablets per day) as needed. They were told not to take any analgesics on the day of follow-up assessments, as this could affect clinical outcome measures.Patients were then questioned about their Paracetamol doses used by the patients at the end of the 1st and 6th months were recorded NRS-11 and WOMAC scores at 1 and 6 months during outpatient clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 40 years of age
* Diagnosed with primary knee osteoarthritis according to ACR (American College of Rheumatology) criteria based on clinical, radiological, and laboratory evaluations
* Activity VAS score of 5 or higher despite previous medical and physical therapy
* Patients with stage 3-4 knee osteoarthritis according to the Kellgren-Lawrence classification
* Patients without motor or sensory loss on neurological examination
* Patients who signed an informed consent form
* Patients who have not undergone any interventional procedures on the knee within the last 6 months

Exclusion Criteria:

* Patients with bleeding or coagulation disorders
* Patients with sepsis or local infection at the intervention site
* Patients with allergies to any of the medications to be used
* Patients without study consent
* Patients with secondary osteoarthritis
* Patients who have undergone knee interventions in the last 6 months
* Patients who have undergone knee surgery
* Psychosis

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who presented to the Algology Clinic of Istanbul Cemil Taşçıoğlu City Hospital with knee pain and were diagnosed with stage 3-4 knee osteoarthritis based on clinical, radiological, and laboratory tests between January 2024 and september 2025 were scheduled for the procedure. The procedure was performed on only one knee; the second knee was not treated.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2025-12-05 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
1. Numeric Rating Scale (NRS-11): The NRS-11 is an 11-point numerical scale (9) that allows patients to rate their pain from 0 (no pain at all) to 10 (the most severe pain they have ever experienced). It was assessed three times: pre-treatment, 1 month a | 6 month

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC): | 6 month
  It is a standardized questionnaire widely used by healthcare professionals to assess the condition of patients with knee and hip osteoarthritis, including pain, stiffness, and physical function of the joints. It was developed in 1982 by Western Ontario and McMaster Universities. Higher scores indicate worse pain, stiffness, and functional limitations. The WOMAC consists of five items for pain (score range 0-20), two items for stiffness (score range 0-8), and 17 items for functional limitations (score range 0-68).

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Küçükçekmece, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided